CLINICAL TRIAL: NCT01598259
Title: Randomized Controlled Trial to Assess Efficacy of Melatonin for Children During Burn Rehabilitation
Acronym: Sleep6
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack or enrollment, funding depletion
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Michele Gottschlich, Research Scientist, Shriners Hospitals for Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-1613
Record Dates: First submitted 2012-05-08; First posted 2012-05-15 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- melatonin (Experimental): Subjects will receive melatonin
  Interventions: Drug: Melatonin
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Melatonin — po 1 hour before bedtime
  Arms: melatonin
Other: placebo — po, 1 hour before bed
  Arms: placebo

SUMMARY:
The specific aims of this investigation in children during burn rehabilitation include 1.) to determine the efficacy of melatonin intervention on improving sleep-related outcomes 2.) investigate the hypothesis that sleep inadequacy is associated with cognitive deficits and 3.) develop a new methodology specific for burn patients that accurately screens for the presence of intrinsic dyssomnia.

ELIGIBILITY:
Inclusion Criteria:

* History of burn injury
* Scheduled for an elective surgical procedure
* 5 - 22 years of age, inclusive

Exclusion Criteria:

* History of anoxic brain injury
* History of head injury within the last year
* Pre-existing seizure disorder
* Pre-existing neurological disorder
* Pre-existing blindness
* Known hypersensitivity to melatonin
* Anticoagulant use or aspirin therapy
* Antihypertensive medication use
* Diabetes mellitus or other endocrine disorders
* Autoimmune disorders
* Schizophrenia
* Inability to access internet
* Intellectual disability or inability to follow directions

Ages: 5 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
sleep | 3 years
  Measure sleep parameters via polysomnography, actigraphy and urinary melatonin

CONTACTS AND LOCATIONS:
Locations (1):
- Shriners Hospital for Children, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
given low level of enrollment and hence, randomization (n=3), no plans to provide data